CLINICAL TRIAL: NCT00703781
Title: Efficacy and Safety of Bromfenac Ophthalmic Solution in Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL-S&E-0415081-P-ER
Record Dates: First submitted 2008-06-20; First posted 2008-06-24 (Estimated); Results first posted 2011-12-09 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Cataract
Keywords: Cataract extraction with intraocular lens implantation
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bromfenac (Experimental): Bromfenac Ophthalmic Solution 0.09%, Dosed 1 Drop Daily
  Interventions: Drug: bromfenac ophthalmic solution
- Placebo (Placebo Comparator): Placebo, Dosed 1 Drop Daily
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: bromfenac ophthalmic solution — sterile ophthalmic solution
  Arms: Bromfenac
Drug: placebo — sterile ophthalmic solution
  Arms: Placebo

SUMMARY:
Efficacy and Safety of Bromfenac Ophthalmic Solution in Cataract Surgery

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for cataract surgery

Exclusion Criteria:

* Known hypersensitivity to bromfenac and salicylates

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- ISTA Pharmaceuticals, Inc., Irvine, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study start date was 06/10/2008 and last participant to exit the study was 09/02/2008. This study was conducted in 18 study centers.
Pre-assignment Details: A total of 126 subjects were randomized to investigational product and were included in the Intent-to-Treat (ITT) population; 63 were randomized to the bromfenac ophthalmic solution treatment group and 63 were randomized to the placebo treatment group.
Period: Overall Study
Arm/Group | Bromfenac | Placebo
Started | 63 | 63
Completed | 61 | 61
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Cancelled surgery | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bromfenac | Placebo | Total
Number analyzed (Participants) | 63 | 63 | 126
Age, Continuous [Mean (Full Range); unit: years] | 67.1 (10.8) [41 to 86] | 68.6 (8.6) [51 to 87] | 67.9 (9.8) [41 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 38 | 78
  Male | 23 | 25 | 48

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Summed Ocular Inflammation Score (SOIS) of Zero
Description: Participants with SOIS of 0. Scale: 0=0 cells (complete absence); 0.5=1-5 cells (trace); 1=6-15 cells (very slight); 2=16-25 cells (moderate); 3=26-50 cells (marked); 4=>50 cells (intense)
Time Frame: Day 15
Population: Last Observation Carried Forward Analysis (LOCF). Intent to treat population (ITT)
Measure: Number; unit: Participants
Arm/Group | Bromfenac | Placebo
Number analyzed (Participants) | 63 | 63
Participants | 28 | 20

2. Secondary Outcome: Number of Participants That Are Pain Free
Description: Participant description of being pain free taken from patient questionnaire with multiple possible responses (None, Mild, Moderate, Severe) within one hour of instilling eye drop
Time Frame: Day 1
Population: LOCF Analysis, ITT Population
Measure: Number; unit: Participants
Arm/Group | Bromfenac | Placebo
Number analyzed (Participants) | 63 | 63
Participants | 51 | 46

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Bromfenac | Placebo
Serious Adverse Events (participants affected / at risk) | 2/61 | 0/61
Other Adverse Events (participants affected / at risk) | 46/61 | 61/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromfenac (N=61) | Placebo (N=61)
Nausea and Vomiting Symptoms (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal Failure (Renal and urinary disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bromfenac (N=61) | Placebo (N=61)
Corneal Edema (Eye disorders) | 4 (4) | 2 (2)
Lacrimation Increased (Eye disorders) | 3 (4) | 6 (7)
Eye Pain (Eye disorders) | 5 (6) | 7 (9)
Eye Inflammation (Eye disorders) | 8 (13) | 14 (15)
Eye Pruritus (Eye disorders) | 6 (6) | 2 (2)
Foreign Body Sensation (Eye disorders) | 8 (8) | 6 (7)
Photophobia (Eye disorders) | 8 (10) | 17 (18)
Vision Blurred (Eye disorders) | 4 (4) | 2 (2)
Ocular Hyperemia (Eye disorders) | 0 (0) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on the PI is that the PI will provide to the sponsor a copy of proposed publication information for review, comment and approval following completion of the study and at least sixty (60) days prior to submission of the publication. If sponsor requests in writing, the PI will withhold publication until written permission is given by sponsor.